CLINICAL TRIAL: NCT02652845
Title: Wellness Engagement Project, Petersburg
Acronym: WE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Design was changed - no longer prospectively assigning participants
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Pathways-VA Inc (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R24MD008128 (NIH); 1R24MD008128 (NIH)
Record Dates: First submitted 2015-06-05; First posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention-Wellness Engagement Program (Experimental): The group assigned to the intervention arm will receive treatment as described below for a twelve week period:
  Weekly lessons related to healthy eating and physical activity Biweekly check-in calls with a trained peer support coach Access to neighborhood wide physical activity and nutritional education events
  Interventions: Behavioral: Wellness Engagement Program
- Delayed treatment control group (No Intervention): The delayed treatment control group will not receive the intervention for measurement purposes; however the intervention as described will be administered to this group upon conclusion of the 12 week period for the intervention group.

INTERVENTIONS:
Behavioral: Wellness Engagement Program — This intervention is an evidence based and community informed program designed to stimulate physical activity and increase healthy food choices among participants. The intervention includes weekly lessons, personal support in the form of biweekly check in calls with a peer support coach and weekly physical activity and nutrition classes.
  Arms: Intervention-Wellness Engagement Program

SUMMARY:
This study tests the feasibility of a health and wellness trial designed with community input. This 12-week program will be tested over a 24-week period using a delayed treatment control group.

DETAILED DESCRIPTION:
This 12-week program was designed based on input from Petersburg, VA community residents, collected through various methods over a two-year period. The 12 week program is designed to impact three levels: individual, family and community. At the individual level, participants receive print material lessons related to healthy eating and increasing physical activity, as well as videos that model these lessons; participants will also have access to a peer support coach who will contact them on a biweekly basis and are trained to help them identify and reach their own personal health goals. At the family level, participants are encouraged to share all of the information they receive as a part of this program with the rest of their family, and are asked to begin walking regularly and to attend fitness and nutrition classes held within their neighborhood (by the WE program) with family members. On a community level, local church groups and neighborhood organizations will receive assistance in launching walking clubs, and all community residents are invited to attend the physical activity and nutrition classes that the WE project hosts within the community.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years.
* Must have a school going child between 12-17 living in the home.
* BMI between 25 and 50 kg/m2.

Exclusion Criteria:

* report not being able to walk 2 blocks (1/4 mile) without stopping
* currently participating in another weight loss program
* taking a weight loss medication
* have a history of bariatric surgery
* pregnant or plan to become pregnant during the intervention timeframe
* report an unsupervised heart condition, chest pain during periods of rest or activity, or loss of consciousness on the Physical Activity Readiness Questionnaire
* report a medical condition that would jeopardize their safety if involved in a weight management program with diet and exercise guidelines (e.g., uncontrolled heart problem)
* fail medical screening by study medical staff)
* report conditions that, in the judgment of the PI, would render the participant unlikely to follow the study protocol (e.g., planned move from the area, dementia, substance abuse).

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Engagement in WE activities | 4-weeks
  Number of community events attended
Video lessons | 4 weeks
  Number of video lessons viewed as reported to Wellness Ambassadors
Peer Support | 4 weeks
  number of check-in phone calls completed with Peer Support Coaches
Self-monitoring logs | 4 weeks
  number of self-monitoring logs completed
Value of the program | 4 weeks
  Perceived value of the program
Effectiveness of peer support | 4 weeks
  Perception of the effectiveness of the peer support received from peer coaches

SECONDARY OUTCOMES:
Uptake of key behaviors promoted in the WE program | 4-weeks
  Engagement in recommended health behaviors
Weight | 4-weeks
  Weight will be measured in kg
Dietary changes | 4-weeks
  Dietary practices will be assessed using the Behavioral Risk Factor Surveillance System (BRFSS)
Height | 4 weeks
  height measured in meters

CONTACTS AND LOCATIONS:
Overall Officials: Maghboeba Mosavel, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States